CLINICAL TRIAL: NCT05473000
Title: Investigating Susceptibility of Cardiorespiratory Responses to Ozone During Cycling Exercise Based on Resting Ozone Exposure
Brief Title: Susceptibility of Cardiorespiratory Responses to Ozone During Cycling Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Michael Koehle, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H22-01389
Record Dates: First submitted 2022-07-12; First posted 2022-07-25 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Ozone Exposure During Rest and Exercise
Keywords: Ozone; Air pollution; Exercise; Cycling; Susceptibility; Ventilation
MeSH Terms: conditions — Motor Activity; Disease Susceptibility; Respiratory Aspiration | interventions — Exercise; Ozone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Air quality (ozone and room air) will be double-blinded; neither participants nor the primary researcher will know the randomized order of the condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone (O3) (Experimental): Participants of the experimental group will perform sub-maximal exercise (power output associated with 10% below anaerobic threshold for 30 minutes) and maximal exercise (time-to-exhaustion test at 5% above previously determined maximal power output) on a cycle ergometer while inhaling 170ppb ozone delivered continuously during each exercise session.
  Interventions: Behavioral: Exercise; Other: Ozone
- Room air (Sham Comparator): Participants of the sham group will perform sub-maximal exercise (power output associated with 10% below anaerobic threshold for 30 minutes) and maximal exercise (time-to-exhaustion test at 5% above previously determined maximal power output) on a cycle ergometer while inhaling room air during each exercise session.
  Interventions: Behavioral: Exercise; Other: Room air

INTERVENTIONS:
Behavioral: Exercise — Submaximal and maximal exercise
Other: Ozone — Delivery of ozone air pollution at 170ppb
  Arms: Ozone (O3)
Other: Room air — Delivery of room air
  Arms: Room air

SUMMARY:
Ground level ozone (O3) is a common airborne pollutant that is well recognized to cause negative respiratory symptoms and impair pulmonary function. The proposed study aims to have participants perform submaximal and maximal cycling exercise protocols exposed to both O3 and room air in a crossover design to evaluate how ventilatory patterns, pulmonary function, development of symptoms, and cycling performance are impacted by O3 exposure. Additionally, the investigators look to compare responses between O3 at rest and during exercise to predict which subjects may be most susceptible to adverse response, as considerable interindividual variability exists.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the age of 18 and 50
* Currently training and/or competing in endurance sport
* VO2max >60 ml/kg/min
* Able to communicate sufficiently using the English language

Exclusion Criteria:

* History of smoking
* Upper respiratory tract infection within the last 4 weeks
* Presence of any chronic respiratory disease

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Koehle, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 participants were screened for inclusion by the researchers during an initial study visit.
Pre-assignment Details: 22 eligible participants were randomized, with 20 opting to complete the two experimental visits in this crossover design.
Groups:
- Ozone (O3) First, Then Room Air: Participants completed submaximal and maximal exercise during a single study visit exposed to O3 (170ppb). After a 72 hour washout period, they then completed identical procedures exposed to room air.
- Room Air First, Then Ozone (O3): Participants completed submaximal and maximal exercise during a single study visit exposed to room air. After a 72 hour washout period, they then completed identical procedures exposed to O3 (170ppb).
Period: First Intervention
Arm/Group | Ozone (O3) First, Then Room Air | Room Air First, Then Ozone (O3)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (Minimum 72 Hours)
Arm/Group | Ozone (O3) First, Then Room Air | Room Air First, Then Ozone (O3)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Ozone (O3) First, Then Room Air | Room Air First, Then Ozone (O3)
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Room Air First, Then Ozone (O3): Participants completed submaximal and maximal exercise during a single study visit exposed to room air. After a 72 hour washout period, they then completed identical procedures exposed to ozone (O3).
- Total: Total of all reporting groups
Arm/Group | Ozone (O3) First, Then Room Air | Room Air First, Then Ozone (O3) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 28 (6) | 28 (6) | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Time-to-exhaustion on Maximal Cycling Bout
Description: Measurement of time (in seconds) to volitional exhaustion on a constant work-rate cycling trial at 110% of previously determined maximal power output.
Time Frame: From the beginning of the maximal constant work-rate cycling bout until volitional exhaustion occurs (roughly 1-5 minutes)
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Ozone (O3): Participants completed submaximal and maximal exercise during a single study visit exposed to O3 (170ppb) during either intervention period.
- Room Air: Participants completed submaximal and maximal exercise during a single study visit exposed to room air during either intervention period.
Arm/Group | Ozone (O3) | Room Air
Number analyzed (Participants) | 19 | 19
seconds | 209 (59) | 235 (81)
Statistical Analysis 1: Comparison: Ozone (O3) vs Room Air; Test type: Superiority; p = 0.092, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the testing period (~4 weeks for participants).
Description: All participants were at risk of adverse events due to exposure to low-levels of air pollution (O3) and maximal exercise.
Groups:
- Ozone (O3): Participants who completed submaximal and maximal exercise during exposure to ozone (O3).
- Room Air: Participants who completed submaximal and maximal exercise during exposure to room air.
Arm/Group | Ozone (O3) | Room Air
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05473000/Prot_SAP_000.pdf